CLINICAL TRIAL: NCT00453232
Title: Accelerated BEP Chemotherapy for Intermediate and High Risk Metastatic Germ Cell Tumor
Brief Title: Combination Chemotherapy and Pegfilgrastim in Treating Men With Metastatic Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CRCA-CCTC-ACCELERATED-BEP; CDR0000537042 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2004-000847-79; EU-20713; ISRCTN18505589 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Extragonadal Germ Cell Tumor; Teratoma; Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; testicular choriocarcinoma and seminoma; testicular embryonal carcinoma and seminoma; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma; testicular choriocarcinoma and yolk sac tumor; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular seminoma; testicular yolk sac tumor; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; recurrent malignant testicular germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; adult teratoma; testicular immature teratoma; testicular mature teratoma; recurrent extragonadal germ cell tumor
MeSH Terms: conditions — Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Carcinoma, Embryonal; Endodermal Sinus Tumor | interventions — Bleomycin; pegfilgrastim; Cisplatin; Etoposide

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: pegfilgrastim
Drug: cisplatin
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bleomycin, etoposide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving combination chemotherapy together with pegfilgrastim may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving combination chemotherapy together with pegfilgrastim works in treating men with metastatic germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of accelerated treatment comprising bleomycin, etoposide, cisplatin, and pegfilgrastim in men with metastatic germ cell tumors.
* Determine the toxicity of this regimen (particularly with respect to renal, pulmonary, and neurological function) in these patients.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.

OUTLINE: This is a non-randomized, pilot study.

Patients receive etoposide IV on days 1-3, cisplatin IV on days 1 and 2, and bleomycin IV over 2 hours on days 2, 6, and 10. Patients also receive pegfilgrastim subcutaneously on day 4. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must fulfill all of the following criteria for 1 of the following diagnoses:

  * Nonseminoma germ cell tumor (intermediate risk)

    * Testis or retroperitoneal primary
    * Abnormal markers (alpha fetoprotein [AFP] > 1,000 and < 10,000 ng/mL, human chorionic gonadotropin [HCG] > 5,000 and < 50,000 IU/L, lactate dehydrogenase [LDH] > 1.5 times and < 10 times upper limit of normal [ULN])
    * No liver, bone, brain, or other nonpulmonary visceral metastasis
    * Histologic confirmation is not required if AFP or HCG are grossly elevated
  * Nonseminoma germ cell tumor (poor prognosis) meeting 1 of the following criteria:

    * Mediastinal primary
    * Nonpulmonary visceral metastases
    * Poor markers (AFP > 10,000 ng/mL, HCG > 50,000 IU/L, LDH > 10 times ULN)
    * Histologic confirmation not required if AFP or HCG are grossly elevated
  * Seminoma (intermediate prognosis)

    * Histological confirmation is required
    * Any primary site
    * Nonpulmonary visceral metastases must be present
    * Normal AFP
    * Any HCG
    * Any LDH
  * Surveillance relapse

    * Must fulfill appropriate criteria above according to initial histology

PATIENT CHARACTERISTICS:

* Neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Must have adequate renal function (creatinine clearance ≥ 60 mL/min)
* No prior malignancy except basal cell carcinoma

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Toxicity
Feasibility

SECONDARY OUTCOMES:
Response rate
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Williams, MD, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Churchill Hospital, Oxford, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland